CLINICAL TRIAL: NCT04569123
Title: Concomitant Sensory Stimulation During Therapy to Enhance Hand Functional Recovery Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro90790; 1R01HD094731-01A1 (NIH)
Record Dates: First submitted 2020-09-23; First posted 2020-09-29 (Actual); Results first posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Physical Disability
Keywords: physical stimulation; subliminal stimulation; stroke rehabilitation; physical therapy; occupational therapy; upper extremity; paresis; hand function
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration (Active Comparator): The device will deliver imperceptible vibration for the treatment group.
  Interventions: Device: real stimulation
- No Vibration (Sham Comparator): The device will deliver no vibration for the control group.
  Interventions: Device: No stimulation

INTERVENTIONS:
Device: real stimulation — Participants will undergo standardized hand task practice therapy (3 sessions/week for 6 weeks) with the watch worn on the paretic wrist. Participants will be randomized into two groups: The device will deliver vibration for the treatment group.
  Arms: Vibration
Device: No stimulation — Participants will undergo standardized hand task practice therapy (3 sessions/week for 6 weeks) with the watch worn on the paretic wrist. Participants will be randomized into two groups: The device will deliver no vibration for the control group during therapy.
  Arms: No Vibration

SUMMARY:
The objective of this study is to determine if combining vibration with hand task practice is superior to hand task practice alone.

DETAILED DESCRIPTION:
Stroke is a leading cause of disability in the U.S., with more than 4 million stroke survivors in the U.S. who suffer from post-stroke hand disability. Post-stroke hand disability impairs stroke survivors' abilities and independence with self-care, hygiene, employment, and leisure, frequently resulting in diminished quality of life. Rehabilitation can often be limited, but research suggests that the effects of therapy is improved by the addition of sensory stimulation.

To fully leverage the potential therapeutic benefits of sensory stimulation, we have developed a new stimulation that is imperceptible random-frequency vibration applied to wrist skin. The objective of this study is to determine if this treatment is superior to task-practice alone in improving hand functional recovery, sensorimotor grip control, and neural communication.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* At least 6 months since stroke
* Wolf Motor Function Test (WMFT) total average time >10 seconds
* WFMT hand task average time <120 s

Exclusion Criteria:

* Currently undergoing other upper limb therapy
* Change in spasticity medication or upper limb botulinum toxin injection within 3 months prior to or during enrollment
* Severe spasticity that limits participation in task practice therapy (e.g., Modified Ashworth Scale=4-5)
* Comorbidity affecting the upper limb function such as complete upper extremity deafferentation, orthopaedic conditions limiting motion, premorbid neurologic conditions, premorbid peripheral neuropathy, compromised skin integrity of the wrist due to burn or long-term use of blood thinners, or significant new neurological symptoms
* Language barrier or cognitive impairment that precludes following instructions and/or providing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-01-06 (Actual); Study Completion 2025-01-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seo NJ, Ramakrishnan V, Woodbury ML, Bonilha L, Finetto C, Schranz C, Scronce G, Coupland K, Blaschke J, Baker A, Howard K, Meinzer C, Velozo CA, Adams RJ. Concomitant sensory stimulation during therapy to enhance hand functional recovery post stroke. Trials. 2022 Apr 5;23(1):262. doi: 10.1186/s13063-022-06241-9. PMID 35382902

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vibration | No Vibration
Started | 30 | 31
Completed | 25 | 22
Not Completed | 5 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vibration | No Vibration | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: year] | 62 (13) | 59 (10) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 14 | 22
  Male | 22 | 17 | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 20 | 30
  White | 19 | 10 | 29
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Wolf Motor Function Test (WMFT) Movement Time
Description: The Wolf Motor Function Test (WMFT) is a standardized, timed assessment of upper extremity motor function. This study reports the total average movement time across the WMFT tasks.
  Range: 0 seconds to >120 seconds (no fixed upper limit). Interpretation: Lower movement times indicate better motor function. Only this WMFT movement-time variable was analyzed as the pre-specified primary outcome.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: Seconds (sec)
Arm/Group | Vibration | No Vibration
Number analyzed (Participants) | 25 | 22
Seconds (sec) | -4 (6) | -9 (10)

2. Secondary Outcome: Change in Box and Blocks Test (BBT) Score
Description: The Box and Blocks Test (BBT) measures unilateral gross manual dexterity. Participants move as many blocks as possible from one side of a box to the other in 60 seconds.
  Range: 0-150 blocks (typical). Interpretation: Higher scores indicate better manual dexterity.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: Number of blocks moved
Arm/Group | Vibration | No Vibration
Number analyzed (Participants) | 25 | 22
Number of blocks moved | 2 (4) | 4 (6)

3. Secondary Outcome: Change in Action Research Arm Test (ARAT) Score
Description: The Action Research Arm Test (ARAT) is a standardized measure of upper limb functional ability. It contains 19 items scored 0-3, summed to a total score.
  Range: 0-57. Interpretation: Higher scores indicate better upper limb function.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Vibration | No Vibration
Number analyzed (Participants) | 25 | 22
Score on a scale | 3 (3) | 4 (5)

ADVERSE EVENTS:
Time Frame: From enrollment through completion of study participation, up to 2.5 months.
Arm/Group | Vibration | No Vibration
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 3/30 | 2/31
Other Adverse Events (participants affected / at risk) | 25/30 | 23/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vibration (N=30) | No Vibration (N=31)
serious adverse event (General disorders) | 3 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vibration (N=30) | No Vibration (N=31)
other adverse event (General disorders) | 25 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT04569123/Prot_SAP_001.pdf
  • Informed Consent Form (2024-08-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT04569123/ICF_000.pdf